CLINICAL TRIAL: NCT02647528
Title: A Randomized, Blinded, Single-Centered, Placebo-Controlled Trial of Pulse Dyed Laser (Chromogenex Regenlite Transform) in the Treatment of Inflammatory Acne Vulgaris
Brief Title: A Trial of Pulse Dyed Laser (Chromogenex Regenlite Transform) in the Treatment of Inflammatory Acne Vulgaris
Acronym: Chromogenix
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: funding withdrawn
Sponsor: Sadick Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Chromogenex Acne
Record Dates: First submitted 2015-12-31; First posted 2016-01-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Patients in this arm receive treatment
  Interventions: Device: Chromogenix Regenlite Transform Treatment
- Placebo (Placebo Comparator): Patients in this arm do not receive treatment
  Interventions: Device: Chromogenix Regenlite Transform Placebo

INTERVENTIONS:
Device: Chromogenix Regenlite Transform Treatment — Pulse Dyed Laser - 7mm spot size 3-3.6 J/cm2
  Arms: Treatment
Device: Chromogenix Regenlite Transform Placebo — Pulse Dyed Laser - 7mm spot size 0 J/cm2
  Arms: Placebo

SUMMARY:
A Randomized, Blinded, Single-Centered, Placebo-Controlled Trial of Pulse Dyed Laser (Chromogenex Regenlite Transform) in the Treatment of Inflammatory Acne Vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained including HIPAA authorization.
* Healthy male or non-pregnant female 18-65 years-of-age with a clinical diagnosis of mild to moderate facial acne vulgaris.
* Subject must have at least eight and not more than fifty inflammatory facial lesions (i.e., papules/pustules) and no nodules on the face. For the purposes of study treatment and evaluation, these lesions should be limited to the facial treatment area including those present on the nose. Lesions involving the eyes, and scalp should be excluded from the count.
* Subject must be in general good health and free from any clinically significant disease, other than acne, that might interfere with the study evaluations.
* Female subjects of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 1 year), in addition to having a negative urine pregnancy test, must be willing to use an acceptable form of birth control during the study from the day of the first dose administration to 30 days after the last administration of study drug.
* Subjects who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to use the same make-up brand/type and frequency of use throughout the study.
* Subjects must agree not to have any other procedures affecting skin quality (microdermabrasion, peels, acne treatments, etc.) for the duration of the study.
* Subjects must understand the study and be able to follow study instructions as well as attend the required study visits.
* Subjects who agree to be photographed for research purposes and their identity may not be concealed in these photographs.

Exclusion Criteria:

* Subjects whom are pregnant, planning to become pregnant or breastfeeding. A urine pregnancy test will be done to rule out pregnancy.
* Subjects of child-bearing potential who are not using an approved method of birth control (oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence). Females of non-childbearing potential are defined as post-menopausal (absence of menstrual bleeding for one year), hysterectomy or bilateral oophorectomy.
* Subjects who cannot understand or are not willing to comply with the requirements of the study.
* Presence of any skin condition on the face that would interfere with the diagnosis or assessment of acne.
* Excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne.
* The use within 6 months prior to baseline of oral retinoids (e.g. Accutane®) or therapeutic vitamin A supplements of greater than 10,000units/day (multivitamins are allowed).
* The use of estrogens or oral contraceptives for less than 3 months prior to baseline.
* The use within 1 month prior to baseline of:

  * topical retinoids to the face;
  * systemic antibiotics known to have an impact on the severity of facial acne (e.g., containing tetracycline and its derivatives, erythromycin and its derivatives, sulfamethoxazole, or trimethoprim);
  * systemic corticosteroids (Note: intranasal and inhalational corticosteroids do not require a washout and maybe used throughout the trial if the subject is on a stable dose).
* Use within 2 weeks prior to baseline of:

  * topical corticosteroids;
  * topical antibiotics;
  * topical medications for acne (e.g., metronidazole).
* Subjects with moderate or severe rhinophyma, dense telangiectases (score 3, severe), or plaque-like facial edema.
* Ocular rosacea (e.g., conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics.
* A subject who has used a sauna during the 2 weeks prior to study entry and during the study.
* Subjects who have performed wax epilation of the face within 14 days prior to baseline.
* A subject with bacterial folliculitis.
* A subject who consumes excessive alcohol, abuses drugs or has a condition that could compromise the subject's ability to comply with study requirements.
* Subjects who engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold.
* A subject who has any clinically significant condition or situation, other than the condition being studied that, in the opinion of the Investigator, would interfere with the study evaluations or optimal participation in the study.
* A subject who has used any topical azelaic acid therapy within 30 days of baseline visit.
* Subjects who have participated in an investigational drug study (i.e., subjects have been treated with an Investigational Drug) within 30 days prior to baseline will be excluded from study participation. Subjects who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion.
* Subjects who have been previously enrolled in this study.
* Subjects who have had laser therapy (for telangiectasia or other conditions), electrodessication and phototherapy to the facial area within 180 days prior to study entry.
* Subjects who have had cosmetic procedures (e.g., facials) which may affect the efficacy and safety profile of the Investigational Product within 14 days prior to study entry.
* Subjects who have had any kind of facial dermabrasion, chemical peel, laser, IPL or any other treatment that could influence the skin quality in the past 6 months or for the duration of the study
* Subjects who do not agree to avoid using tanning beds or intensive exposure to the sun two weeks prior to each office visit.
* Subjects who have any known cancer including skin cancers (basal cell carcinoma, squamous cell carcinoma and melanoma) in the treatment area.
* Subjects who are currently involved in any injury litigation claims.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Global Acne Assessment Scoring | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sadick Research Group, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No